CLINICAL TRIAL: NCT05648968
Title: A Phase 3, Randomized, Double-blind, Study to Assess Efficacy and Safety of Ianalumab (VAY736) Versus Placebo in Warm Autoimmune Hemolytic Anemia (wAIHA) Patients Who Failed at Least One Line of Treatment
Brief Title: A Study of Efficacy and Safety of Ianalumab in Previously Treated Patients With Warm Autoimmune Hemolytic Anemia
Acronym: VAYHIA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736O12301; 2022-001773-31 (EudraCT Number); 2024-510635-21-00 (Other: EMA (EU CTR ID))
Expanded Access: NCT07244289 (Available)
Record Dates: First submitted 2022-11-23; First posted 2022-12-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Warm Autoimmune Hemolytic Anemia (wAIHA)
Keywords: warm autoimmune hemolytic anemia; wAIHA; ianalumab; VAY736; B-cell depletion; B-cell Activating Factor Receptor (BAFF-R) blockade
MeSH Terms: interventions — ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ianalumab low dose (Experimental): Participants will receive low dose ianalumab intravenously
  Interventions: Biological: Ianalumab
- Ianalumab high dose (Experimental): Participants will receive high dose ianalumab intravenously
  Interventions: Biological: Ianalumab
- Placebo (Placebo Comparator): Participants will receive placebo intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Ianalumab — i.v. infusion, prepared from concentrate solution
  Other Names: VAY736
  Arms: Ianalumab high dose; Ianalumab low dose
Drug: Placebo — i.v. infusion, prepared from matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of ianalumab compared to placebo in patients with warm autoimmune hemolytic anemia, who failed at least one line of treatment.

DETAILED DESCRIPTION:
The primary objective is to demonstrate that either dose of ianalumab induces a durable hemoglobin response compared to placebo in patients with wAIHA.

The key secondary objective is to demonstrate that either dose of ianalumab maintains a durable hemoglobin response that is sustained beyond end of the treatment period, compared to placebo.

Participants are randomized to two different doses of ianalumab or placebo. Participants who were assigned to placebo arm and not responding to treatment may be treated with open label ianalumab using the higher dose.

The investigational treatment will be supplied in a double-blinded manner. For the open label period, ianalumab will be provided in an open label manner.

In addition to the randomized treatment (ianalumab or placebo), specific supportive care medication as defined in the protocol is allowed. If clinically indicated (e.g., to ensure patient safety), the treating physician may also administer rescue medication.

The study consists of the treatment period, efficacy and safety follow-up periods. The visit frequency will be every other week during the treatment and primary endpoint follow up period; for safety monitoring monthly during the first 20 weeks after last dose and afterwards quarterly up to 2 years from the last dose. For participants in durable response, additional visits for efficacy will occur monthly during the first 2 years after the last dose, and afterwards quarterly until loss of response or end of study, latest until up to 39 months post randomization of the last participant.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 years and older at time of signing consent
* Patients with primary or secondary wAIHA documented by positive direct antiglobulin test specific for anti-IgG or anti-IgA, who had an insufficient response to, or relapsed after at least one line of treatment, including patients with steroid resistance, dependence or intolerance
* Hemoglobin concentration at screening and at Week 1 >=5 g/dL and <10 g/dL, associated with presence of symptoms related to anemia
* The dose of supportive care must be stable for at least 4 weeks prior to randomization into the study

Key Exclusion Criteria:

* wAIHA secondary to hematologic disease involving bone marrow (e.g., CLL) or another immunologic disease requiring prohibited medication as per protocol. Patients with autoimmune diseases after wash-out from the treatments are allowed.
* Presence of other forms of AIHA (cold or intermediate forms), Evans Syndrome or other cytopenias
* Prior use of B-cell depleting therapy (e.g., rituximab) within 12 weeks prior to randomization, or without hematological response to the last course of B-cell depleting therapy
* Neutrophils: <1000/mm3
* Serum creatinine >1.5 × upper limit of normal (ULN)
* Immunoglobulin G (IgG) <5g/L
* Active viral, bacterial or other infections (including tuberculosis and SARS-CoV-2) requiring systemic treatment at time of screening, or history of recurrent clinically significant infection
* Positivity for hepatitis C virus, hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb). HBcAb positive patients can be enrolled if HBsAg negative, HBV DNA negative, no pre-existing liver fibrosis is present and antiviral prophylaxis is given.
* Known history of primary or secondary immunodeficiency, or a positive human immune deficiency virus (HIV) test result
* Live or live-attenuated vaccination within 4 weeks before randomization
* History of splenectomy

Other protocol-defined Inclusion/Exclusion may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2028-12-19 (Estimated)

PRIMARY OUTCOMES:
Binary variable indicating whether a patient achieves a durable response | Randomization to Week 25
  Durable response: hemoglobin level ≥10 g/dL and ≥2 g/dL increase from baseline, for a period of at least eight consecutive weeks between W9 and W25, in the absence of rescue medication or prohibited treatment

SECONDARY OUTCOMES:
Duration of response (Key Secondary) | Randomization to end of study (up to 39 months after randomization of last patient)
  • For patients who previously reached durable response:
  Time from first hemoglobin assessment showing durable response to confirmed loss of durable response, defined as the first of the following events:
  * hemoglobin level <10 g/dL in at least two consecutive weekly assessments,
  * start of any rescue medication or prohibited treatment,
  * death; • For patients who did not achieve the durable response according to primary endpoint definition: duration will be 0 days
Time from randomization to start of durable response in each treatment group | Randomization to end of study (up to 39 months after randomization of last patient)
  Durable response is defined as in primary endpoint.
Time from randomization to start of first response in each treatment group | Randomization to end of study (up to 39 months after randomization of last patient)
  Response is defined as hemoglobin level of at least 10 g/dL and an increase of at least 2 g/dl from baseline, or normalization of hemoglobin (at least 11 g/dL for women and 12 g/dL for men), without biochemical resolution of hemolysis.
Time from randomization to start of complete response in each treatment group | Randomization to end of study (up to 39 months after randomization of last patient)
  Complete response is defined as normalization of hemoglobin levels and no evidence of hemolysis (normal levels of indirect bilirubin, LDH, haptoglobin and reticulocytes), in the absence of red blood cell transfusions.
Response rate | Randomization to end of study (up to 39 months after randomization of last patient)
  Assessment of quality of response in each treatment group.
Complete response rate | Randomization to end of study (up to 39 months after randomization of last patient)
  Assessment of complete response rate in each treatment group.
Hemoglobine Levels | Randomization to end of study (up to 39 months after randomization of last patient)
  Assessment of hemoglobin levels in each treatment group.
Number of participants who received rescue treatment (overall & by type of rescue treatment) | Randomization to end of study (up to 39 months after randomization of last patient)
  This is to assess the need for rescue treatment in all treatment groups, measured as time-standardized numbers of each type of rescue treatment and as change from baseline in time-standardized number of transfusions.
Percentage of participants who received rescue treatment (overall & by type of rescue treatment) | Randomization to end of study (up to 39 months after randomization of last patient)
  This is to assess the need for rescue treatment in all treatment groups.
Change from baseline in the the frequency and absolute number of CD19+ B cell counts | Randomization to end of study (up to 39 months after randomization of last patient)
  Change from baseline in the the frequency and absolute number of CD19+ B cell counts in whole blood
Time to first occurrence of B cell recovery, defined as ≥80% of baseline or ≥50 cells/μL | Randomization to end of study (up to 39 months after randomization of last patient)
  Time to first occurrence of B cell recovery, defined as ≥80% of baseline or ≥50 cells/μL in whole blood
Change from baseline in immunoglobulin levels | Randomization until month 30
  Change from baseline in immunoglobulin levels (change in titers of IgG, IgM, IgA)
Change from baseline in the 8 domain scores and in the summary scores (PCS, MCS) of SF-36 questionnaire | Randomization to end of study (up to 39 months after randomization of last patient)
  SF-36 v2.0 (acute) includes 36 items that assess general health related quality of life covering 8 domains: physical functioning, role functioning, bodily pain, general health, vitality, social functioning, role-emotional health and mental health.
  Scores for the 8 domains are generated, as well as a physical component summary (PCS) score and a mental component summary (MCS) score.
  Responses to items are based on a 5-point Likert scale. Scores below 50 indicate less than average health, while scores above 50 indicate better than average health.
Change from baseline in the T-score of PROMIS Fatigue-13a questionnaire | Randomization to end of study (up to 39 months after randomization of last patient)
  Assessment of quality of life in each treatment group. The PROMIS Short Form v1.0 Fatigue-13a includes 13 items that assess fatigue. All items in the PROMIS-Fatigue-13a utilize a 5-point response scale (e.g., not at all, a little bit, somewhat, quite a bit, very much).
  Higher scores on the PROMIS-Fatigue-13a represent greater fatigue.
Ianalumab PK parameter - AUClast | After first dose of study treatment (pre-dose, 2 hours, 336 hours, 672 hours post dose) and after last dose (pre-dose, 2 hours, 336 hours, 672 hours, 1344 hours, 2016 hours and 3360 hours post dose).
  AUClast: area under the curve from time zero to last measurable concentration sampling time (tlast).
Ianalumab PK parameter - AUCtau | After first dose of study treatment (pre-dose, 2 hours, 336 hours, 672 hours post dose) and after last dose (pre-dose, 2 hours, 336 hours, 672 hours, 1344 hours, 2016 hours and 3360 hours post dose).
  AUCtau: the AUV calculated to the end of a dosing interval (tau).
Ianalumab PK parameter - Accumulation ratio Racc | After last dose (pre-dose, 2 hours, 336 hours, 672 hours, 1344 hours, 2016 hours and 3360 hours post dose).
  Accumulation ratio calculated using AUC values obtained between last and first dose
Ianalumab PK parameter - Cmax | After first dose of study treatment (pre-dose, 2 hours, 336 hours, 672 hours post dose) and after last dose (pre-dose, 2 hours, 336 hours, 672 hours, 1344 hours, 2016 hours and 3360 hours post dose).
  Maximum (peak) observed plasma, blood, serum or other body fluid drug concentration
Ianalumab PK parameter - Tmax | After first dose of study treatment (pre-dose, 2 hours, 336 hours, 672 hours post dose) and after last dose (pre-dose, 2 hours, 336 hours, 672 hours, 1344 hours, 2016 hours and 3360 hours post dose).
  Time to reach maximum (peak) plasma, blood, serum or other body fluid drug concentration
Immunogenicity of ianalumab | Randomization to end of study (up to 39 months after randomization of last patient)
  Incidence and titer of anti-ianalumab antibodies in serum (ADA assay) over time. Confirmed anti-drug-antibody positive samples will be further characterized for neutralizing capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (51):
- United States (4):
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - University of Minnesota Med Center, Minneapolis, Minnesota
  - Summit Health, Florham Park, New Jersey
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Argentina (2):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Caba
- Australia (3):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
- China (4):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Dalian
  - Novartis Investigative Site, Tianjin
- France (5):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Toulouse
- Germany (4):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Hanover
- Novartis Investigative Site, Debrecen, Hajdu Bihar Megye, Hungary
- India (4):
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
- Israel (2):
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Bassano del Grappa, VI
  - Novartis Investigative Site, Novara
- Japan (8):
  - Novartis Investigative Site, Narita, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
- Malaysia (3):
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Johor Bahru
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Murcia
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- United Kingdom (3):
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com